CLINICAL TRIAL: NCT01016054
Title: A Phase 1b, Parallel Arm, Multicenter, Open-Label Study of the Safety and Pharmacokinetics of AGS-8M4 Given in Combination With Two Different Chemotherapy Regimens in Women With Platinum Resistant or Platinum Sensitive Ovarian Cancer
Brief Title: A Study of the Safety and Pharmacokinetics of AGS-8M4 Given in Combination With Chemotherapy in Women With Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was terminated to allow sponsors to evaluate the future development of the drug program
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009001
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Carcinoma; Ovarian Cancer; Ovarian Diseases; Ovarian Neoplasms
Keywords: Clinical Trial, Phase1; Combination Drug Therapy; pharmacokinetics; safety; Ovarian
MeSH Terms: conditions — Carcinoma; Ovarian Neoplasms; Ovarian Diseases | interventions — liposomal doxorubicin; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. PLD plus AGS-8M4 (Experimental): Women with platinum resistent ovarian cancer
  Interventions: Biological: AGS-8M4; Drug: Pegylated liposomal doxorubicin (PLD)
- B. Carboplatin and gemcitabine plus AGS-8M4 (Experimental): Women with platinum sensitive ovarian cancer
  Interventions: Biological: AGS-8M4; Drug: gemcitabine; Drug: carboplatin

INTERVENTIONS:
Biological: AGS-8M4 — IV infusion
Drug: Pegylated liposomal doxorubicin (PLD) — IV infusion
  Arms: A. PLD plus AGS-8M4
Drug: gemcitabine — IV infusion
  Arms: B. Carboplatin and gemcitabine plus AGS-8M4
Drug: carboplatin — IV infusion
  Arms: B. Carboplatin and gemcitabine plus AGS-8M4

SUMMARY:
This is a parallel arm study to evaluate AGS-8M4 administered in combination with chemotherapy in subjects with ovarian cancer. AGS-8M4 will be administered as an IV infusion until disease worsens.

DETAILED DESCRIPTION:
All Subjects will receive AGS-8M4 treatment. Subjects will be enrolled into 1 of 2 treatment arms according to their disease status. A disease assessment will be performed every 8 or 9 weeks (± 3 days) depending on the treatment arm assignment. The assessment will be based both on changes in clinical symptoms, and radiographic images. Subjects without evidence of disease progression may continue to receive treatment based on their original treatment assignment until disease progression or intolerability. A safety follow-up visit will occur 4 weeks after the last dose infusion of AGS-8M4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with recurrent disease Stage III/IV diagnosis of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma
* Subjects with either platinum resistant or platinum sensitive ovarian cancer
* At least 14 days of previous cytotoxic chemotherapy and have recovered from all toxicities
* Left ventricular ejection fraction (LVEF) equal to or greater than the institutional lower limit of normal as measured by echocardiogram or MUGA (ONLY required for platinum resistant patients)

Exclusion Criteria:

* Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) within 72 hours of screening
* Use of any investigational drug within 30 days prior to screening
* Prior monoclonal antibody therapy other than Avastin
* Avastin administration within 90 days of screening
* History of thromboembolic events and bleeding disorders ≤ 3 months (e.g.,DVT or PE)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Throughout the treatment

SECONDARY OUTCOMES:
Assessment of PK variables | Treatment Arm A: Weeks 1 and 3 of each cycle. Treatment Arm B: Week 1 of each cycle. In addition, samples will be drawn at the Safety F/U, 2 Month F/U and 3 Month F/U visits.
Incidence of anti-AGS-8M4 antibody formation | Treatment Arm A: Day 1 of every other cycle and at Day 15 for the first cycle only. Treatment Arm B: Day 1 of every other cycle. In addition, samples will be drawn at the Safety F/U, 2 Month F/U and 3 Month F/U visits.
Changes in tumor status per RECIST | Treatment Arm A: Every 8 weeks. Treatment Arm B: Every 9 weeks.
Change in CA-125 levels | Treatment Arm A: Day 1 and Day 15 of each cycle. Treatment Arm B: Day 1 of each cycle. In addition, samples will be drawn at the Safety F/U.

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Agensys, Inc.
Locations (1):
- Duarte, California, United States